CLINICAL TRIAL: NCT04579055
Title: The Impact of Chair Seat Height on the 1-Minute Sit to Stand Test Performance in Chronic Obstructive Pulmonary Disease: a Randomized Cross-over Study
Brief Title: Impact of Chair Seat Height on the 1-Minute Sit to Stand Test Performance in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Riegler (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Thomas Riegler, Principal Investigator, Berner Reha Zentrum AG
Organization: Berner Reha Zentrum AG (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2020-01677
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease
Keywords: 1-minute Sit to Stand Test; chair seat height
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-min STS test: chair seat height adjusted to 90° knee flexion (Experimental): In this experimental condition, the patient performs the 1-minute sit to stand test on an individually adjusted seat height of 90° knee joint flexion.
  Interventions: Other: 1-min STS test: adjusted
- 1-min STS test: chair seat height standardized of 46cm (Active Comparator): In this experimental condition, the patient performs the 1-minute sit to stand test on a standard height chair of 46cm.
  Interventions: Other: 1-min STS test: standardized

INTERVENTIONS:
Other: 1-min STS test: adjusted — Individually adjusted chair seat height of 90° knee joint flexion
  Arms: 1-min STS test: chair seat height adjusted to 90° knee flexion
Other: 1-min STS test: standardized — Standardized chair seat height of 46 cm
  Arms: 1-min STS test: chair seat height standardized of 46cm

SUMMARY:
The 1-minute sit to stand (1-min STS) test is a standardized test which is used to examine exercise capacity in patients with chronic obstructive pulmonary disease (COPD). The chair seat height used is standardized to 46-48 cm. Using a standard seat height for all patients - irrespective of their body height - may lead to invalid estimates of functional exercise capacity. The objective of this study is to assess whether there is a difference in repetitions during the 1-min STS test if the seat height is adjusted to 90° knee joint angle or the standard height chair of 46 cm is used.

DETAILED DESCRIPTION:
In a single-center, randomized crossover study, the investigators aim to elucidate whether there is a difference in repetitions during the 1-min STS test if the seat height is adjusted to 90° knee joint angle or the standard height chair of 46 cm is used.

Patients with COPD referred for pulmonary rehabilitation will be invited to perform one standardised- (chair seat height 46cm) and one individualized (chair seat height adapted to 90° knee flexion) 1-min STS test on two different days in random order.

The tests will be performed after patients are familiarised with the 1-min STS testing procedure and learning effects can be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed COPD according to a forced expiratory volume in 1s (FEV1) / forced vital capacity (FVC) ratio below the lower limit of normal

Exclusion Criteria:

* Patients who are not able to bend their knees while sitting on a standard chair (i.e., knee flexion less than 90°)
* Patients who are not able to understand the instructions of the 1-min STS test, either of language or cognitive reasons
* Patients who are unable to perform the STS test due to functional disability (i.e., being not able to rise from a chair without hand support), previous surgery, or pain according to the judgement of the responsible physician.
* Patients who did not sign the informed consent form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Number of repetitions in the 1-min STS test | During pulmonary rehabilitation, approximately 14 days
  difference in the amount of sit to stand repetitions in the 1-min STS test from a standard chair (46cm) or an individualized seat height chair of 90° knee joint angle

SECONDARY OUTCOMES:
Sit to stand power index | During pulmonary rehabilitation, approximately 14 days
  The sit to stand power index is used to calculate the force-generating capacity (in watt) of the knee extensor muscles and is defined as: (leg length (in m) - seat height (in m)) x body mass x acceleration of gravity x sit to stand repetitions / time (sit-stand) (in sec.)

OTHER OUTCOMES:
Oxygen saturation | During pulmonary rehabilitation, approximately 14 days
  Difference in oxygen saturation profiles between the two experimental conditions
Heart rate | During pulmonary rehabilitation, approximately 14 days
  Difference in heart rate profiles between the two experimental conditions
Ratings of perceived exertion | During pulmonary rehabilitation, approximately 14 days
  Difference in perceived exertion profiles between the two experimental conditions measured with the category ratio - 10 Borg scale (0-10)
Ratings of perceived breathlessness | During pulmonary rehabilitation, approximately 14 days
  Difference in perceived breathlessness profiles between the two experimental conditions measured with the category ratio - 10 Borg scale (0-10)
Incorrectly performed repetitions during the 1-min STS test | During pulmonary rehabilitation, approximately 14 days
  The number of incorrectly performed repetitions during th 1-min STS test
Questionnaire about the patient's preferences during the 1-min sit to stand test | During pulmonary rehabilitation, approximately 14 days
  Multiple choice questions about patient reported perception concerning sitting position, chair height, perceived difficulties during the 1-min sit to stand test.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Riegler, MSc, Principal Investigator — Berner Reha Zentrum, Heiligenschwendi; Thomas Radtke, PD, Dr phil, Principal Investigator — University of Zurich
Locations (1):
- Berner Reha Zentrum, Heiligenschwendi, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crook S, Busching G, Schultz K, Lehbert N, Jelusic D, Keusch S, Wittmann M, Schuler M, Radtke T, Frey M, Turk A, Puhan MA, Frei A. A multicentre validation of the 1-min sit-to-stand test in patients with COPD. Eur Respir J. 2017 Mar 2;49(3):1601871. doi: 10.1183/13993003.01871-2016. Print 2017 Mar. PMID 28254766
- [Background] Yoshioka S, Nagano A, Hay DC, Fukashiro S. Peak hip and knee joint moments during a sit-to-stand movement are invariant to the change of seat height within the range of low to normal seat height. Biomed Eng Online. 2014 Mar 12;13(1):27. doi: 10.1186/1475-925X-13-27. PMID 24620992
- [Background] Reychler G, Boucard E, Peran L, Pichon R, Le Ber-Moy C, Ouksel H, Liistro G, Chambellan A, Beaumont M. One minute sit-to-stand test is an alternative to 6MWT to measure functional exercise performance in COPD patients. Clin Respir J. 2018 Mar;12(3):1247-1256. doi: 10.1111/crj.12658. Epub 2017 Jun 15. PMID 28621019
- [Background] Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, Enright PL, Hankinson JL, Ip MS, Zheng J, Stocks J; ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012 Dec;40(6):1324-43. doi: 10.1183/09031936.00080312. Epub 2012 Jun 27. PMID 22743675
- [Background] Miller MR, Quanjer PH, Swanney MP, Ruppel G, Enright PL. Interpreting lung function data using 80% predicted and fixed thresholds misclassifies more than 20% of patients. Chest. 2011 Jan;139(1):52-9. doi: 10.1378/chest.10-0189. Epub 2010 Jun 3. PMID 20522571